CLINICAL TRIAL: NCT05834595
Title: An Open-label, Randomized, Fasted, Single-dose, 2-sequence, 4-period, Replicate Crossover Study to Compare the Pharmacokinetic and Safety Between Administration of CKD-828 20/2.5mg and Administration of D064, D701 in Healthy Adults
Brief Title: A Clinical Trial to Compare the Pharmacokinetic and Safety of CKD-828
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A30_19BE2305
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: D064, D701 - A single oral dose of 2 tablets
  * Period 2: CKD-828 - A single oral dose of 1 tablet
  * Period 3: D064, D701 - A single oral dose of 2 tablets
  * Period 4: CKD-828 - A single oral dose of 1 tablet
  Interventions: Drug: CKD-828, D064, D701
- Sequence 2 (Experimental): * Period 1: CKD-828 - A single oral dose of 1 tablet
  * Period 2: D064, D701 - A single oral dose of 2 tablets
  * Period 3: CKD-828 - A single oral dose of 1 tablet
  * Period 4: D064, D701 - A single oral dose of 2 tablets
  Interventions: Drug: CKD-828, D064, D701

INTERVENTIONS:
Drug: CKD-828, D064, D701 — QD, PO

SUMMARY:
A clinical trial to compare the pharmacokinetic and safety of CKD-828

DETAILED DESCRIPTION:
An open-label, randomized, fasted, single-dose, 2-sequence, 4-period, replicate crossover study to compare the pharmacokinetic characteristics and safety between administration of CKD-828 20/2.5mg and administration of D064, D701 in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged ≥ 19 at screening
2. Body mass index (BMI) of 17.5 kg/m2 or more and less than 30.5kg/m2 and Body weight ≥ 55kg
3. Those who do not have congenital or chronic diseases and have no pathological symptoms or findings as a result of medical examination
4. A person who is deemed suitable as a subject as a result of screening such as clinical laboratory examination (hematology, blood chemistry, urinalysis, serological tests, etc.), vital signs, electrocardiogram examination, etc.
5. A person who has received a sufficient explanation of the purpose and contents of the clinical trial and has agreed in writing voluntarily to participate in the clinical trial
6. A person who has agreed to use appropriate contraception and not donate sperm or eggs until 14 days after the first administration of the drug and the last administration of the drug
7. Those who have the ability and willingness to participate during the entire study period

Exclusion Criteria:

1. A history of clinically significant blood, renal, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, psychiatric, neurological, or immune disease (except for simple dental history of calculus, impacted teeth, wisdom teeth, etc.) or evidence on who has
2. Those with a history of gastrointestinal diseases or surgery (expect simple appendicectomy, hernia surgery, and tooth extraction surgery) that may affect drug absorption ruler
3. A person who shows the following values as a result of conducting a clinical laboratory test

   * ALT or AST > 2 times the upper limit of the normal range
4. Smokers who smoked more than 20 cigarettes a day within 6 months of screening
5. Those who have taken other investigational product or bioequivalence investigational product within 6 months before the first administration of the investigational product
6. Those who meet the following as a result of measuring vital signs at screening

   * Those who have a systolic blood pressure of less than 90 mmHg or more than 140 mmHg or a diastolic blood pressure of less than 60 mmHg or more than 90 mmHg in the sitting position
   * Severe bradycardia (less than 50 beats/min)
7. Those with a history of regular alcohol intake within 1 month of screening

   * More than 14 drinks/week for women
   * More than 21 drinks/week for men
8. A person who has taken a drug known to significantly induce or inhibit drug metabolizing enzymes within 30 days before the first administration of investigational product
9. Those who have taken prescription or non-prescription drugs within 10 days prior to the first administration of investigational product
10. Those who have donated whole blood within 2 months before the first administration of the investigational product, donated component blood within 1 month, received blood transfusion within 1 month, or have plans for the trial during the clinical trial period
11. Those who are judged by the principal investigator (or the person in charge of the test who has been delegated) for reason other than the above selection/exclusion criteria and are judged unsuitable for participation in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-828 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72 hours
  Area under the concentration-time curve time zero to time
Cmax of CKD-828 | Pre-dose(0 hour), 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 48, 72 hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Central hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No